CLINICAL TRIAL: NCT00424255
Title: A Randomised, Double-Blind, Placebo-Controlled, Multi-centre, Phase III Study of Post-Operative Adjuvant Lapatinib or Placebo and Concurrent Chemoradiotherapy Followed by Maintenance Lapatinib or Placebo Monotherapy in High-Risk Subjects With Resected Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Study Of Adjuvant Lapatinib In High-Risk Head And Neck Cancer Subjects After Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EGF102988
Record Dates: First submitted 2007-01-17; First posted 2007-01-19 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-06

CONDITIONS: Neoplasms, Head and Neck
Keywords: Cancer of the Head and Neck; Neck cancer; Adjuvant; Head and neck cancer; High-risk head and neck cancer; Post-surgery; Head cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Lapatinib; Chemoradiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Lapatinib+Chemoradiation (Experimental): Adjuvant concurrent chemoradiotherapy plus lapatinib 1500 mg once daily for 6 to 7 weeks, followed by lapatinib 1500 mg once daily for one year.
  Chemoradiotherapy=total dose of 66Gy over 6-7 weeks plus cisplatin 100mg/m2 on days 1,2 and 43 of the course of radiotherapy. Lapatinib is also given at 1500 mg once daily for 3-7 days prior to the start of chemoradiotherapy.
  Interventions: Drug: Lapatinib
- Placebo+Chemoradiation (Placebo Comparator): Adjuvant concurrent chemoradiotherapy plus placebo once daily for 6 to 7 weeks, followed by placebo once daily for one year.
  Chemoradiotherapy = total dose of 66Gy over 6-7 weeks plus cisplatin 100mg/m2 on days 1,2 and 43 of the course of treatment. Placebo is also given once daily for 3-7 days prior to the start of chemoradiotherapy.
  Interventions: Radiation: Chemoradiation; Other: Placebo

INTERVENTIONS:
Drug: Lapatinib — Dual ErbB1/2 inhibitor
  Arms: Lapatinib+Chemoradiation
Radiation: Chemoradiation — Radiation plus platinum based chemotherapy
  Arms: Placebo+Chemoradiation
Other: Placebo — Placebo
  Arms: Placebo+Chemoradiation

SUMMARY:
This is a randomised, double-blind, placebo-controlled, multicentre, global Phase III trial comparing the efficacy of adjuvant oral lapatinib versus placebo in high-risk subjects with head and neck cancer following surgery. Lapatinib or placebo will be administered post-operatively in combination with chemoradiotherapy followed by maintenance with lapatinib or placebo for 1 year. The primary goal is to determine if lapatinib is effective at reducing the recurrence of the disease in these high-risk patients.

DETAILED DESCRIPTION:
A Randomised, Double-Blind, Placebo-Controlled, Multi-centre, Phase III Study of Post-Operative Adjuvant Lapatinib or Placebo and Concurrent Chemoradiotherapy Followed by Maintenance Lapatinib or Placebo Monotherapy in High-Risk Subjects with Resected Squamous Cell Carcinoma of the Head and Neck (SCCHN)

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign a written informed consent.
* Histologically confirmed diagnosis of SCCHN of one of the following sites: oral cavity, oropharynx, hypopharynx and larynx.
* Pathological Stage II, III or IVa (according to AJCC cancer staging criteria [Green, 2002]) with no evidence of gross residual disease, and at least one of the following high risk factors by pathology:
* Extracapsular extension of nodal disease
* Positive resection margin (5 mm or less)
* Primary surgery with a curative intent completed within 4-6 weeks (and no later than 7 weeks) prior to randomization. The extent of surgical resection will follow accepted criteria for adequate excision [Helliwell, 2005]. Surgical margins are divided into 'mucosal' and 'deep', and for each category the resection margin (R) is classified as:
* Clear : (R0) > 5mm.
* Close: (R1) 1 - 5mm.
* Involved: (R2) <1mm
* Complete recovery from the surgical procedure allowing for appropriate radiotherapy. Radiation therapy is required to start as soon as adequate healing has occurred. This is normally around 4-6 weeks but no later than 9 weeks after surgery.
* Adequate tumour specimen from archived or resected tissue must be available for IHC evaluation of ErbB1 expression levels in a central laboratory and subsequent biomarker analysis.
* Male or female, between 18 and 70 years of age [Bourhis, 2006].

Criteria for female subjects or female partners of male subjects:

Non-child-bearing potential (i.e., a woman with functioning ovaries who has a current documented tubal ligation or hysterectomy or a woman who is menopausal); or

Child-bearing potential (i.e. a woman with functioning ovaries and no documented impairment of oviductal or uterine function that would cause sterility. This category includes women with oligomenorrhoea (even severe), women who are perimenopausal and young women who have begun to menstruate), who have a negative serum pregnancy test at screening, and agree to one of the following:

Complete abstinence from intercourse from the time of the screening pregnancy test until 28 days after the final dose of test article; or

Consistent and correct use of one of the following acceptable methods of birth control:

Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject; or Oral contraceptives (either combined or progestogen only), or Injectable progestogen-only contraceptives or Implants of levonorgestrel, or Any intrauterine device with a documented failure rate of less than 1% per year; or Barrier methods (e.g. condoms, diaphragms, caps) only if used in combination with one of the above acceptable methods.

* ECOG performance status 0, 1 or 2
* Adequate haematology, renal and hepatic function Absolute neutrophil count ≥ 1,500/μL, platelets ≥ 100,000/μL Haemoglobin ≥ 9 gm/dL (5mmol/L) Calculated creatinine clearance ≥60 ml/min as determined by the modified method of Cockcroft and Gault.

Aspartate (AST) and alanine transaminase (ALT) less than 3 times the upper limit of the normal range (ULN).

Total bilirubin ≤ 2.0 mg/dL

* Left ventricular ejection fraction (LVEF) above the lower limits of the institutional normal range as measured by ECHO (if ECHO cannot be performed or if the Investigator feels it is not conclusive to evaluate LVEF, then a MUGA scan should be performed).
* Able to swallow and retain tablets whole or swallow a suspension of tablets dissolved in water at study inclusion.

The use of feeding tube is optional. If necessary, the suspension may be administered via percutaneous endoscopic gastrostomy (PEG), percutaneous jejunostomy tube (J- Tube), or a nasogastric tube (NG or Dobhoff type tube).

* Life expectancy of at least 6 months in the best judgement of the investigator
* Current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, or stable chronic liver disease per investigator assessment).

Exclusion Criteria:

* Nasopharyngeal, paranasal sinuses or nasal cavity tumours
* Head and neck cancer with histology other than squamous cell carcinoma.
* Evidence of distant metastases or gross post-operative residual disease.
* Evidence of second primary tumour.
* Any prior or current anticancer treatment of any kind - except the primary surgical resection. This will include but is not limited to: prior tyrosine kinase inhibitors, prior neoadjuvant therapy, prior radiotherapy or use of any investigational agent.
* Concurrent treatment with an investigational agent or participation in another clinical trial.
* Concurrent use of CYP3A4 inducers or inhibitors while on lapatinib/placebo. A standard 3 to 5 day course of dexamethasone for the prevention of cisplatin induced nausea and vomiting is permitted. In addition glucocorticoid daily doses (oral) 1.5mg dexamethasone (or equivalent) are allowed.
* Subjects with known history of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure;
* Pregnant or lactating females
* History of another malignancy within the last 5 years, with the exception of completely resected basal or squamous cell skin cancer, or successfully treated in-situ carcinoma. History of non-invasive lesion or in-situ carcinoma, that was successfully treated with surgery, photodynamics or laser, will be permitted;
* Peripheral neuropathy ≥ grade 2
* Mal-absorption syndrome, disease significantly affecting GI function, or major resection of the stomach or bowel, that could affect absorption of lapatinib.
* History of allergic reactions to relevant diuretics or anti-emetics (e.g 5-HT3 antagonists) to be administered with cisplatin chemotherapy
* History of allergic reactions attributed to compounds of similar chemical composition (quinazolines) to lapatinib
* The investigator considers the subject unfit for the study as a result of the medical interview, physical examinations, or screening investigations

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Actual)
Dates: Start 2006-12; Primary Completion 2013-03 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (101):
- United States (5):
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Lubbock, Texas
- Argentina (4):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Santa Fe, Santa Fe Province
  - GSK Investigational Site, Quilmes
- Austria (4):
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Rankweil
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Vienna
- Canada (5):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- China (6):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Fuzhou
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin
- GSK Investigational Site, Zagreb, Croatia
- Czechia (4):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Prague
- GSK Investigational Site, Tallinn, Estonia
- France (15):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Annecy
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Colmar
  - GSK Investigational Site, Férolles-Attilly
  - GSK Investigational Site, La Roche-sur-Yon
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Reims
  - GSK Investigational Site, Saint-Cloud
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Villejuif
- Germany (6):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Karlsruhe, Baden-Wurttemberg
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Halle, Saxony-Anhalt
- Greece (4):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Haidari, Athens
  - GSK Investigational Site, Neo Faliro
  - GSK Investigational Site, Peiraius
- Hong Kong (2):
  - GSK Investigational Site, Hong Kong
  - GSK Investigational Site, Kowloon
- Hungary (2):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Szombathely
- India (4):
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Trivandrum
- Ireland (2):
  - GSK Investigational Site, Galway
  - GSK Investigational Site, Rathgar, Dublin
- Italy (5):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Venezia, Veneto
- GSK Investigational Site, Manila, Philippines
- Russia (3):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Ufa
- Slovakia (2):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
- Spain (14):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Huesca
  - GSK Investigational Site, Lleida
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Ourense
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Zaragoza
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
- United Kingdom (9):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Northwood, Middlesex
  - GSK Investigational Site, Edinburgh, Midlothian
  - GSK Investigational Site, Brighton, Sussex East
  - GSK Investigational Site, Guildford
  - GSK Investigational Site, London
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Sheffield
  - GSK Investigational Site, Sutton

REFERENCES:
- [Derived] Sunkara PR, Chow E, Waitzman J, Sukari A, Cramer JD. The Prognostication of Surgically Resected Head and Neck Squamous Cell Carcinoma Using Pre-Therapy Neutrophil and Lymphocyte Counts. Head Neck. 2025 Feb;47(2):687-694. doi: 10.1002/hed.27949. Epub 2024 Oct 16. PMID 39415507
- [Derived] Sunkara PR, Graff JT, Cramer JD. Association of Surgical Margin Distance With Survival in Patients With Resected Head and Neck Squamous Cell Carcinoma: A Secondary Analysis of a Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2023 Apr 1;149(4):317-326. doi: 10.1001/jamaoto.2022.5186. PMID 36821132
- [Derived] Harrington K, Temam S, Mehanna H, D'Cruz A, Jain M, D'Onofrio I, Manikhas G, Horvath Z, Sun Y, Dietzsch S, Dubinsky P, Holeckova P, El-Hariry I, Franklin N, Biswas-Baldwin N, Legenne P, Wissel P, Netherway T, Farrell J, Ellis C, Wang-Silvanto J, Amonkar M, Ahmed N, Santillana S, Bourhis J. Postoperative Adjuvant Lapatinib and Concurrent Chemoradiotherapy Followed by Maintenance Lapatinib Monotherapy in High-Risk Patients With Resected Squamous Cell Carcinoma of the Head and Neck: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study. J Clin Oncol. 2015 Dec 10;33(35):4202-9. doi: 10.1200/JCO.2015.61.4370. Epub 2015 Nov 2. PMID 26527790

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo per oral monotherapy once daily (QD) for 1 week, followed by radiotherapy of 2 Gray (Gy) per day for 5 days per week (for a total dose of 66 Gy for up to 7 weeks). Participants received concurrent cisplatin 100 milligrams per meters squared (mg/m^2) intravenously (IV) on Days 1, 22, and 43 of radiotherapy. One week prior to the start of chemoradiotherapy, then concurrently for 6 to approximately 7 weeks with chemoradiotherapy, participants received placebo per oral administration QD, followed by maintenance placebo per oral monotherapy QD for up to 1 year or until evidence of disease relapse, whichever was sooner.
- Lapatinib 1500 mg: Participants received lapatinib 1500 mg per oral monotherapy QD for 1 week, followed by radiotherapy of 2 Gy per day for 5 days per week (for a total of 66 Gy for up to 7 weeks). Participants received concurrent cisplatin 100 mg/m^2 IV on Days 1, 22, and 43 of radiotherapy. One week prior to the start of chemoradiotherapy, then concurrently for 6 to approximately 7 weeks with chemoradiotherapy, participants received lapatinib 1500 mg per oral administration QD, followed by maintenance lapatinib 1500 mg per oral monotherapy QD for up to 1 year or until evidence of disease relapse, whichever was sooner.
Period: Overall Study
Arm/Group | Placebo | Lapatinib 1500 mg
Started | 342 | 346
Completed | 0 | 0
Not Completed | 342 | 346
Not completed — Death | 115 | 111
Not completed — Lost to Follow-up | 26 | 20
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 34 | 38
Not completed — Physician Decision | 3 | 7
Not completed — Cognitive Disturbance | 1 | 0
Not completed — Non-compliance by Participants | 1 | 0
Not completed — Fatigue | 1 | 0
Not completed — Disease Progression | 0 | 2
Not completed — Sponsor Terminated Study | 161 | 167

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lapatinib 1500 mg | Total
Number analyzed (Participants) | 342 | 346 | 688
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.7 (9.85) | 53.8 (8.38) | 53.8 (9.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 60 | 115
  Male | 287 | 286 | 573
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 1 | 0 | 1
  Asian - Central/South Asian Heritage | 61 | 53 | 114
  Asian - East Asian Heritage | 41 | 47 | 88
  Asian - South East Asian Heritage | 19 | 23 | 42
  Asian - Mixed Race | 0 | 1 | 1
  White - Arabic/North African Heritage | 1 | 3 | 4
  White - White/Caucasian/European Heritage | 219 | 219 | 438

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS)
Description: DFS is defined as the time from randomization until the earliest date of disease recurrence (evidence of local, regional, or distant disease progression, second primary tumor) or death due to any cause. Disease recurrence was based on the assessments from the blinded, independent reviewer (radiological and clinical). Participants who initiated alternative anti-cancer therapy prior to disease recurrence or death were treated as censored at the last assessment prior to the time of this initiation. For participants whose disease did not recur or who did not die, DFS was censored at the time of the last independently assessed radiological scan (where initiation of alternative anti-cancer therapy had not commenced). Participants who missed two or more consecutive disease assessments were censored at the last assessment prior to the missed assessments. Participants considered to have malignant disease at Baseline were censored at the time of randomization.
Time Frame: From randomization until the earliest date of disease recurrence or death due to any cause (average of 101 study weeks)
Population: Intent-to-Treat (ITT) Population: all participants who were randomized to study treatment, irrespective of whether they actually received study medication
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 342 | 346
Months | NA [54.6 to NA] — Because of an insufficient number of events, the median and the upper limit of the confidence interval were not reached. | 53.6 [45.8 to NA] — Because of an insufficient number of events, the upper limit of the confidence interval was not reached.
Statistical Analysis 1: Comparison: Placebo vs Lapatinib 1500 mg; Test type: Superiority or Other; p = 0.2251, Non-stratified log-rank test — The one-sided p-value is unstratified as there are too few events per stratum to perform a stratified test
Statistical Analysis 2: Comparison: Placebo vs Lapatinib 1500 mg; Test type: Superiority or Other; p = 0.4502, Non-stratified log-rank test — The two-sided p-value is unstratified as there are too few events per stratum to perform a stratified test
Statistical Analysis 3: Comparison: Placebo vs Lapatinib 1500 mg; Test type: Superiority or Other; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.85 to 1.43] — Hazard Ratios were estimated using a Pike estimator

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization until death due to any cause. For participants who did not die, the time to death was censored at the time of last visit/contact.
Time Frame: From randomization until death due to any cause (average of 131 study weeks)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 342 | 346
Months | NA [NA to NA] — Because of an insufficient number of events, the median and the upper limit of the confidence interval were not reached. | NA [58.8 to NA] — Because of an insufficient number of events, the median and the confidence intervals were not reached.

3. Secondary Outcome: Disease Specific Survival (DSS)
Description: DSS is defined as the time from randomization until death due to head and neck cancer. Participants whose death was not related to the disease under study were treated as competing risks at the time death occured. Participants who were alive were censored at the time of their last visit.
Time Frame: From randomization until death due to head and neck cancer (average of 131 study weeks)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 342 | 346
Months | NA [NA to NA] — Because of an insufficient number of events, the median and the confidence interval were not reached. | NA [NA to NA] — Because of an insufficient number of events, the median and the confidence interval were not reached.

4. Secondary Outcome: Time to Locoregional Recurrence (TTLR)
Description: TTLR is defined as the time from randomization until the first occurrence that local and/or regional recurrence is documented or the date of censor. Local relapse is defined as recurrent cancer in the primary tumor bed not clearly attributable to a second primary neoplasm. Regional relapse is defined as recurrent cancer in the neck not clearly attributable to a second primary neoplasm. All other events prior to locoregional recurrence were treated as competing risks at the time they occured. All other participants were treated as censored at the time of their last disease assessment. Participants with malignant disease at Baseline according to the independent review were censored at the time of randomization for the analysis of independently reviewed data.
Time Frame: From randomization until thefirst occurrence that local and/or regional recurrence is documented or the date of censor (average of 101 study weeks)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 342 | 346
Months | NA [NA to NA] — Because of an insufficient number of events, the median and confidence interval were not reached. | NA [NA to NA] — Because of an insufficient number of events, the median and the confidence interval were not reached.

5. Secondary Outcome: Time to Distant Relapse (TTDR)
Description: TTDR is defined as the time from randomization until the first occurrence that distant relapse is documented. Distant relapse is defined as clear evidence of distant metastases (lung, bone, brain, etc.). Metastasis is defined as the spread of a cancer from one organ or part to another non-adjacent organ or part. All other events prior to a distant relapse were treated as competing risks at the time they occured. All other participants were treated as censored at the time of their last disease assessment. Participants with malignant disease at Baseline according to the independent review were censored at the time of randomization for the analysis of independently reviewed data.
Time Frame: From randomization until the first documented occurrence that distant relapse is documented (average of 101 study weeks)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 342 | 346
Months | NA [NA to NA] — Because of an insufficient number of events, the median and confidence interval were not reached. | NA [NA to NA] — Because of an insufficient number of events, the median and confidence interval were not reached.

6. Secondary Outcome: Number of Participants With a Second Primary Tumor
Description: Participants who developed a second primary tumor at the time of the first recurrence or within 28 days of the first recurrence were measured. The criteria for a second primary tumor are as follows: a distinct lesion separated from the primary tumor site by >2 centimeters of normal epithelium; or a new cancer with different histology; or any cancer, regardless of site, occurring >=3 years after initial treatment. Participants with baseline disease were included in the denominator when calculating the percentage.
Time Frame: From randomization until development of second primary tumor or within 28 days of first recurrence (average of 101 study weeks)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 342 | 346
Participants | 5 | 9

7. Secondary Outcome: Extent of Exposure
Description: Extent of exposure is defined as the duration of treatment administered during the study. The mean duration of treatment is calculated as the number of days between the start of treatment and the end of treatment inclusive (i.e., treatment stop date minus treatment start date + 1). Participants were counted in a treatment phase (monotherapy, chemoradiotherapy, and maintenance) if they had received any dose in that phase. Participants randomized to placebo who received >=1 dose of lapatinib in error were included in the lapatinib arm.
Time Frame: From randomization until end of 1year maintenance treatment (average of 63 study weeks)
Population: Safety Population (SP): all participants (par.) who were randomized and took >=1 dose of study medication. Only par. available at the specified time points were analyzed (represented by n=X, X in the category titles). Different par. may have been analyzed for different parameters, so the overall number of par. analyzed reflects everyone in the SP.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 336 | 349
Weeks
  Monotherapy, n=332, 347 | 0.9 (0.32) | 0.9 (0.27)
  Chemoradiotherapy, n=327, 344 | 6.6 (1.29) | 6.5 (1.58)
  Maintenance, n=309, 321 | 41.5 (20.00) | 41.1 (21.03)

8. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. Medical or scientific judgment should be exercised in deciding whether reporting is appropriate in other situations. Refer to the General Adverse AE/SAE module for a complete list of non-serious AEs occurring at a frequency threshold of 5% and SAEs.
Time Frame: From the first dose of lapatinib/placebo until 5 days after the last dose (average of 141 study weeks)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 336 | 349
Participants
  Any AE | 328 | 344
  Any SAE | 133 | 169

9. Secondary Outcome: Number of Participants With the Indicated Chemistry Toxicities by Maximum Toxicity Grade (G3 and G4) at the Worst-case On-therapy Visit
Description: Data are summarized using the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 3 (NCI CTC version 3.0) toxicity grades. Data are reported as the number of participants who had a grade 3 (G3) or grade 4 (G4) toxicity for the indicated chemistry parameters, where G3 indicates a severe toxicity and G4 indicates a life-threatening toxicity. Clinical chemistry parameters included: albumin, alkaline phosphatase (AP), alanine amino transferase (ALT), aspartate amino transeferase (AST), total bilirubin (TB), calcium, carbon dioxide content/bicarbonate (CO2/HCO3), creatinine, glucose, potassium, and sodium. The worst-case on-therapy visit includes any scheduled or unscheduled post-Baseline visit.
Time Frame: From Baseline (within 8 weeks prior to randomization [Day 1]) until the end of the maintenance period/early withdrawal (up to Study Week 64)
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the Safety Population.
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 336 | 349
Participants
  Albumin, Grade 3, n=330, 343 | 1 | 0
  Albumin, Grade 4, n=330, 343 | 0 | 0
  AP, Grade 3, n=333, 347 | 1 | 2
  AP, Grade 4, n=333, 347 | 0 | 0
  ALT, Grade 3, n=333, 348 | 9 | 3
  ALT, Grade 4, n=333, 348 | 1 | 0
  AST, Grade 3, n=333, 347 | 5 | 5
  AST, Grade 4, n=333, 347 | 1 | 0
  TB, Grade 3, n=333, 348 | 3 | 6
  TB, Grade 4, n=333, 348 | 0 | 0
  Hypercalcemia , Grade 3, n=333, 348 | 3 | 1
  Hypercalcemia , Grade 4, n=333, 348 | 1 | 1
  Hypocalcemia , Grade 3, n=333, 348 | 1 | 7
  Hypocalcemia , Grade 4, n=333, 348 | 1 | 3
  CO2/HCO3, Grade 3, n=187, 207 | 0 | 1
  CO2/HCO3, Grade 4, n=187, 207 | 0 | 0
  Creatinine, Grade 3, n=333, 348 | 3 | 9
  Creatinine, Grade 4, n=333, 348 | 2 | 0
  Hyperglycemia, Grade 3, n=332, 344 | 6 | 8
  Hypergylcemia, Grade 4, n=332, 344 | 1 | 0
  Hypoglycemia, Grade 3, n=332, 344 | 1 | 1
  Hypogylcemia, Grade 4, n=332, 344 | 2 | 2
  Hyperkalemia, Grade 3, n=333, 348 | 5 | 8
  Hyperkalemia, Grade 4, n=333, 348 | 2 | 2
  Hypokalemia, Grade 3, n=333, 348 | 17 | 35
  Hypokalemia, Grade 4, n=333, 348 | 1 | 7
  Hypernatremia, Grade 3, n=333, 348 | 0 | 0
  Hypernatremia, Grade 4, n=333, 348 | 1 | 1
  Hyponatremia, Grade 3, n=333, 348 | 59 | 85
  Hyponatremia, Grade 4, n=333, 348 | 11 | 0

10. Secondary Outcome: Number of Participants With the Indicated Hematological Toxicities by Maximum Toxicity Grade (G3 and G4) at the Worst-case On-therapy Visit
Description: Data are summarized using the NCI CTC version 3.0 toxicity grades. Data are reported as the number of participants who had a grade 3 (G3) or grade 4 (G4) toxicity for the indicated hematological parameters, where G3 indicates a severe toxicity and G4 indicates a life-threatening toxicity. The worst-case on-therapy visit includes any scheduled or unscheduled post-Baseline visit. Hematology parameter included: hemoglobin, total neutrophils (TN), platelet count (PC), and White Blood Cell (WBC) count.
Time Frame: From Baseline (within 8 weeks prior torandomization [Day 1]) until the end of the maintenance period/early withdrawal (up to Study Week 64)
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 336 | 349
Participants
  Hemoglobin, Grade 3, n=333, 348 | 10 | 13
  Hemoglobin, Grade 4, n=333, 348 | 0 | 3
  Lymphocytes, Grade 3, n=333, 348 | 203 | 208
  Lymphocytes, Grade 4, n=333, 348 | 34 | 48
  TN, Grade 3, n=333, 348 | 57 | 47
  TN, Grade 4, n=333, 348 | 6 | 13
  PC, Grade 3, n=333, 348 | 0 | 3
  PC, Grade 4, n=333, 348 | 2 | 2
  WBC, Grade 3, n=333, 348 | 70 | 72
  WBC, Grade 4, n=333, 348 | 3 | 6

11. Secondary Outcome: Number of Participants With On-therapy and Follow-up Late Radiation Morbidity Events
Description: Late radiation morbidity event data are summarized as the number of participants with late radiation morbidity events per system organ class (SOC). Late radiation effects are defined as those that first occur 90 days or more after the initiation of radiation therapy.
Time Frame: From 180 days after completion of radiation until the last follow-up/withdrawal visit (average of 64 study weeks)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 336 | 349
Participants
  Gastrointestinal disorders | 25 | 23
  General disorders | 8 | 13
  Skin and subcutaneous tissue disorders | 8 | 13
  Musculoskeletal and connective tissue | 13 | 6
  Respiratory, thoracic and mediastinal | 10 | 7
  Injury, poisoning and procedural | 13 | 3
  Nervous system disorders | 6 | 8
  Endocrine disorders | 4 | 3
  Infections and infestations | 3 | 4
  Investigations | 3 | 3
  Vascular disorders | 4 | 2
  Blood and lymphatic system disorders | 2 | 1
  Ear and labyrinth disorders | 2 | 1
  Metabolism and nutrition disorders | 0 | 1
  Neoplasm benign, malignant and unspecified | 1 | 0

12. Secondary Outcome: Change From Baseline in Blood Pressure at the Indicated Time Points
Description: Blood pressure measurement included systolic blood pressure (SBP) and diastolic blood pressure (DBP) at Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, End of CRT, MW 8, MW 16, MW 24, MW 32, MW 40, MW 48, MW 56, and at the time of withdrawal from IP. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, End of chemoradiotherapy (CRT), Maintenance Week (MW) 8, MW 16, MW 24, MW 32, MW 40, MW 48, MW 56, Withdrawal from investigational product (IP; up to Study Week 64)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 336 | 349
Millimeters of mercury (mmHg)
  SBP, Week 1, n=312, 339 | -0.29 (14.153) | 1.24 (14.273)
  SBP, Week 2, n=303, 327 | -2.40 (13.815) | -1.56 (16.415)
  SBP, Week 3, n=310, 319 | -2.64 (14.784) | -1.62 (15.046)
  SBP, Week 4, n=312, 319 | -4.32 (15.414) | -2.63 (17.044)
  SBP, Week 5, n=302, 303 | -4.05 (15.490) | -3.09 (16.472)
  SBP, Week 6, n=307, 307 | -4.70 (15.571) | -4.07 (15.726)
  SBP, Week 7, n=282, 289 | -4.06 (14.774) | -4.86 (17.046)
  SBP, End of CRT, n=304, 310 | -4.79 (15.216) | -4.69 (16.692)
  SBP, MW 8, n=280, 279 | -2.80 (14.137) | -3.58 (15.030)
  SBP, MW 16, n=257, 270 | -2.86 (15.251) | -2.44 (15.718)
  SBP, MW 24, n=234, 252 | -3.44 (15.918) | -2.48 (15.793)
  SBP, MW 32, n=212, 237 | -1.71 (14.936) | -2.55 (15.470)
  SBP, MW 40, n=202, 222 | -1.76 (14.979) | -1.84 (17.358)
  SBP, MW 48, n=199, 210 | -1.57 (15.531) | -1.79 (15.700)
  SBP, MW 56, n=188, 204 | -1.53 (13.942) | -1.64 (15.878)
  SBP, Withdrawal from IP, n=99, 84 | -2.54 (15.746) | -1.38 (17.895)
  DBP, Week 1, n=312, 339 | -0.07 (9.214) | 0.63 (9.719)
  DBP, Week 2, n=303, 327 | -0.81 (8.690) | -0.24 (9.933)
  DBP, Week 3, n=310, 319 | -0.46 (9.245) | -0.68 (9.704)
  DBP, Week 4, n=312, 319 | -2.54 (9.929) | -2.03 (9.797)
  DBP, Week 5, n=302, 303 | -1.38 (10.100) | -1.60 (9.679)
  DBP, Week 6, n=307, 307 | -1.85 (10.673) | -2.37 (9.514)
  DBP, Week 7, n=282, 289 | -1.73 (11.095) | -2.93 (9.402)
  DBP, End of CRT, n=304, 310 | -1.97 (10.224) | -2.11 (10.117)
  DBP, MW 8, n=280, 279 | -0.80 (9.598) | -1.17 (9.877)
  DBP, MW 16, n=257, 270 | -0.36 (9.980) | -0.98 (9.527)
  DBP, MW 24, n=234, 252 | -1.26 (9.956) | -1.65 (9.842)
  DBP, MW 32, n=212, 237 | -0.38 (9.677) | -1.34 (9.929)
  DBP, MW 40, n=202, 222 | -0.69 (9.809) | -0.69 (11.540)
  DBP, MW 48, n=199, 210 | 0.34 (10.797) | -0.56 (10.057)
  DBP, MW 56, n=188, 204 | 0.20 (9.721) | -0.47 (10.475)
  DBP, Withdrawal from IP, n=99, 84 | -0.27 (10.256) | -0.85 (11.806)

13. Secondary Outcome: Change From Baseline in Heart Rate at the Indicated Time Points
Description: Heart rate (HR) was measured at Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, End of CRT, MW 8, MW 16, MW 24, MW 32, MW 40, MW 48, MW 56, and at the time of withdrawal from IP. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, End of chemoradiotherapy (CRT), Maintenance Week (MW) 8, MW 16, MW 24, MW 32, MW 40, MW 48, MW 56, Withdrawal from IP (up to Study Week 64)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 336 | 349
Beats per minute
  Week 1, n=312, 337 | -0.18 (10.414) | -0.84 (10.710)
  Week 2, n=303, 326 | -0.99 (10.910) | -1.17 (10.258)
  Week 3, n=306, 319 | -0.45 (10.701) | -1.24 (9.766)
  Week 4, n=307, 318 | -0.86 (11.116) | -0.39 (11.645)
  Week 5, n=298, 303 | -0.68 (11.673) | -0.39 (11.588)
  Week 6, n=306, 306 | -0.73 (11.933) | -0.43 (10.947)
  Week 7, n=279, 288 | 1.22 (11.491) | 0.40 (11.184)
  End of CRT, n=300, 310 | 0.33 (12.362) | 0.54 (11.683)
  MW 8, n=279, 277 | -0.30 (10.684) | 0.85 (10.632)
  MW 16, n=256, 268 | -1.10 (11.238) | -0.96 (11.129)
  MW 24, n=235, 251 | -0.98 (11.180) | -1.16 (9.793)
  MW 32, n=213, 238 | -1.43 (11.934) | -1.24 (10.549)
  MW 40, n=203, 222 | -2.72 (11.781) | -0.96 (10.556)
  MW 48, n=200, 210 | -2.56 (12.158) | -0.93 (11.659)
  MW 56, n=189, 204 | -3.08 (12.056) | -1.16 (11.331)
  Withdrawal from IP, n=99, 83 | 0.02 (12.719) | -0.69 (11.822)

14. Secondary Outcome: Change From Baseline in Body Temperature at the Indicated Time Points
Description: Body temperature was measured at Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, End of CRT, MW 8, MW 16, MW 24, MW 32, MW 40, MW 48, MW 56, and at the time of withdrawal from IP. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: as for outcome 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Degrees Centigrade
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 336 | 349
Degrees Centigrade
  Week 1, n=308, 331 | -0.03 (0.420) | -0.01 (0.436)
  Week 2, n=303, 321 | -0.01 (0.492) | 0.01 (0.410)
  Week 3, n=308, 315 | 0.02 (0.504) | 0.01 (0.431)
  Week 4, n=306, 317 | 0.02 (0.511) | 0.04 (0.494)
  Week 5, n=300, 303 | -0.00 (0.514) | 0.03 (0.416)
  Week 6, n=301, 302 | 0.06 (0.586) | 0.02 (0.540)
  Week 7, n=277, 288 | 0.02 (0.526) | 0.06 (0.507)
  End of CRT, n=297, 305 | 0.04 (0.545) | 0.03 (0.469)
  MW 8, n=274, 273 | 0.02 (0.529) | 0.01 (0.442)
  MW 16, n=253, 263 | -0.02 (0.525) | -0.03 (0.400)
  MW 24, n=227, 244 | -0.03 (0.516) | 0.04 (0.425)
  MW 32, n=207, 235 | -0.04 (0.559) | -0.02 (0.453)
  MW 40, n=199, 219 | -0.04 (0.542) | -0.00 (0.429)
  MW 48, n=195, 205 | -0.02 (0.645) | -0.01 (0.464)
  MW 56, n=184, 200 | -0.01 (0.563) | -0.02 (0.466)
  Withdrawal from IP, n=97, 78 | 0.00 (0.562) | 0.03 (0.419)

15. Secondary Outcome: Change From Baseline in Body Weight at the Indicated Time Points
Description: Body weight was measured at Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, End of CRT, MW 8, MW 16, MW 24, MW 32, MW 40, MW 48, MW 56, and at the time of withdrawal from IP. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: as for outcome 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 336 | 349
Kilograms
  Week 1, n=317, 343 | 0.28 (2.301) | -0.04 (2.263)
  Week 2, n=314, 336 | -0.39 (2.320) | -0.90 (2.747)
  Week 3, n=319, 328 | -1.01 (2.638) | -1.46 (2.889)
  Week 4, n=316, 324 | -1.74 (3.116) | -2.24 (3.352)
  Week 5, n=307, 309 | -2.46 (3.424) | -3.30 (3.803)
  Week 6, n=314, 307 | -3.22 (3.868) | -4.15 (3.912)
  Week 7, n=290, 297 | -4.21 (4.072) | -4.94 (4.266)
  End of CRT, n=309, 311 | -4.54 (4.566) | -5.36 (4.406)
  MW 8, n=287, 287 | -4.56 (5.851) | -5.67 (5.326)
  MW 16, n=257, 275 | -4.31 (6.521) | -5.64 (6.120)
  MW 24, n=236, 252 | -4.26 (7.251) | -5.15 (6.723)
  MW 32, n=220, 241 | -4.17 (7.685) | -4.73 (6.711)
  MW 40, n=208, 224 | -3.63 (7.889) | -4.24 (7.348)
  MW 48, n=197, 212 | -3.20 (7.951) | -3.44 (7.087)
  MW 56, n=191, 206 | -2.95 (8.427) | -3.47 (7.440)
  Withdrawal from IP, n=106, 86 | -4.21 (6.785) | -4.81 (7.649)

16. Secondary Outcome: Number of Participants With Abnormal 12-lead Electrocardiogram (ECG) Findings at the Indicated Time Points
Description: A 12-lead ECG was recorded at Baseline, at the end of the CRT, at Maintenance Week 56, at withdrawal from IP, and at anytime post-baseline. Data are presented as clinically significant (CS) or not clinically significant (NCS) abnormal findings. The study investigator determined if an abnormal ECG finding was CS or NCS.
Time Frame: Baseline (BL; within 8 weeks prior to randomization [Day 1]), End of CRT, Maintenance Week 56, Withdrawal from IP, and at any time Post-Baseline (up to Study Week 64)
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 336 | 349
Participants
  BL, Abnormal NCS, n=334, 349 | 82 | 78
  BL, Abnormal CS, n=334, 349 | 1 | 0
  End of CRT, Abnormal NCS, n=287, 292 | 76 | 71
  End of CRT, Abnormal CS, n=287, 292 | 2 | 2
  Maintenance Week 56, Abnormal NCS, n=166, 174 | 32 | 32
  Maintenance Week 56, Abnormal CS, n=166, 174 | 2 | 0
  Withdrawal from IP, Abnormal NCS, n=70, 59 | 16 | 12
  Withdrawal from IP, Abnormal CS, n=70, 59 | 1 | 1
  Anytime post-baseline, Abnormal NCS, n=307, 312 | 94 | 88
  Anytime post-baseline, Abnormal CS, n=307, 312 | 4 | 3

17. Secondary Outcome: Number of Participants With the Indicated Eastern Cooperative Oncology Group (ECOG) Performance Status Value
Description: The Eastern Cooperative Oncology Group (ECOG) performance status scales and grades/criteria are used by doctors and researchers to assess how a participant's disease is progressing, to assess how the disease affects the daily living abilities of the participant, and to determine appropriate treatment and prognosis. Grade 0, fully active, able to carry on all pre-disease performance without restriction. Grade 1, restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. Grade 2, ambulatory and capable of all selfcare, but unable to carry out any work activities; up and about more than 50% of waking hours. Grade 3, capable of only limited selfcare; confined to bed or chair more than 50% of waking hours. Grade 4, completely disabled; cannot carry on any selfcare; totally confined to bed or chair. Grade 5, dead.
Time Frame: From Baseline (BL; within 8 weeks prior to randomization [Day 1]) until the end of the maintenance period/early withdrawal (up to Study Week 64)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 336 | 349
Participants
  BL, ECOG 0, n=336, 349 | 173 | 179
  BL, ECOG 1, n=336, 349 | 161 | 157
  BL, ECOG 2, n=336, 349 | 2 | 13
  Week 1, ECOG 0, n=319, 342 | 160 | 174
  Week 1, ECOG 1, n=319, 342 | 156 | 159
  Week 1, ECOG 2, n=319, 342 | 3 | 9
  Week 1, ECOG 3, n=319, 342 | 0 | 0
  Week 1, ECOG 4-5, n=319, 342 | 0 | 0
  Week 2, ECOG 0, n=313, 333 | 142 | 149
  Week 2, ECOG 1, n=313, 333 | 166 | 168
  Week 2, ECOG 2, n=313, 333 | 5 | 16
  Week 2, ECOG 3, n=313, 333 | 0 | 0
  Week 2, ECOG 4-5, n=313, 333 | 0 | 0
  Week 3, ECOG 0, n=310, 329 | 138 | 131
  Week 3, ECOG 1, n=310, 329 | 169 | 183
  Week 3, ECOG 2, n=310, 329 | 3 | 15
  Week 3, ECOG 3, n=310, 329 | 0 | 0
  Week 3, ECOG 4-5, n=310, 329 | 0 | 0
  Week 4, ECOG 0, n=317, 327 | 115 | 111
  Week 4, ECOG 1, n=317, 327 | 191 | 194
  Week 4, ECOG 2, n=317, 327 | 11 | 21
  Week 4, ECOG 3, n=317, 327 | 0 | 1
  Week 4, ECOG 4-5, n=317, 327 | 0 | 0
  Week 5, ECOG 0, n=307, 312 | 100 | 95
  Week 5, ECOG 1, n=307, 312 | 191 | 183
  Week 5, ECOG 2, n=307, 312 | 16 | 30
  Week 5, ECOG 3, n=307, 312 | 0 | 4
  Week 5, ECOG 4-5, n=307, 312 | 0 | 0
  Week 6, ECOG 0, n=312, 309 | 97 | 88
  Week 6, ECOG 1, n=312, 309 | 187 | 186
  Week 6, ECOG 2, n=312, 309 | 26 | 32
  Week 6, ECOG 3, n=312, 309 | 2 | 3
  Week 6, ECOG 4-5, n=312, 309 | 0 | 0
  Week 7, ECOG 0, n=284, 295 | 83 | 88
  Week 7, ECOG 1, n=284, 295 | 175 | 176
  Week 7, ECOG 2, n=284, 295 | 23 | 30
  Week 7, ECOG 3, n=284, 295 | 3 | 1
  Week 7, ECOG 4-5, n=284, 295 | 0 | 0
  End of CRT, ECOG 0, n=307, 315 | 95 | 84
  End of CRT, ECOG 1, n=307, 315 | 184 | 186
  End of CRT, ECOG 2, n=307, 315 | 25 | 45
  End of CRT, ECOG 3, n=307, 315 | 3 | 0
  End of CRT, ECOG 4-5, n=307, 315 | 0 | 0
  Maintenance week 8, ECOG 0, n=286, 290 | 132 | 128
  Maintenance week 8, ECOG 1, n=286, 290 | 146 | 153
  Maintenance week 8, ECOG 2, n=286, 290 | 7 | 9
  Maintenance week 8, ECOG 3, n=286, 290 | 1 | 0
  Maintenance week 8, ECOG 4-5, n=286, 290 | 0 | 0
  Maintenance week 16, ECOG 0, n=260, 273 | 135 | 129
  Maintenance week 16, ECOG 1, n=260, 273 | 124 | 138
  Maintenance week 16, ECOG 2, n=260, 273 | 1 | 6
  Maintenance week 16, ECOG 3, n=260, 273 | 0 | 0
  Maintenance week 16, ECOG 4-5, n=260, 273 | 0 | 0
  Maintenance week 24, ECOG 0, n=235, 251 | 122 | 127
  Maintenance week 24, ECOG 1, n=235, 251 | 110 | 119
  Maintenance week 24, ECOG 2, n=235, 251 | 3 | 5
  Maintenance week 24, ECOG 3, n=235, 251 | 0 | 0
  Maintenance week 24, ECOG 4-5, n=235, 251 | 0 | 0
  Maintenance week 32, ECOG 0, n=218, 241 | 117 | 123
  Maintenance week 32, ECOG 1, n=218, 241 | 99 | 115
  Maintenance week 32, ECOG 2, n=218, 241 | 2 | 1
  Maintenance week 32, ECOG 3, n=218, 241 | 0 | 2
  Maintenance week 32, ECOG 4-5, n=218, 241 | 0 | 0
  Maintenance week 40, ECOG 0, n=208, 227 | 118 | 130
  Maintenance week 40, ECOG 1, n=208, 227 | 88 | 94
  Maintenance week 40, ECOG 2, n=208, 227 | 2 | 2
  Maintenance week 40, ECOG 3, n=208, 227 | 0 | 1
  Maintenance week 40, ECOG 4-5, n=208, 227 | 0 | 0
  Maintenance week 48, ECOG 0, n=205, 214 | 121 | 111
  Maintenance week 48, ECOG 1, n=205, 214 | 81 | 102
  Maintenance week 48, ECOG 2, n=205, 214 | 3 | 1
  Maintenance week 48, ECOG 3, n=205, 214 | 0 | 0
  Maintenance week 48, ECOG 4-5, n=205, 214 | 0 | 0
  Maintenance week 56, ECOG 0, n=194, 211 | 107 | 111
  Maintenance week 56, ECOG 1, n=194, 211 | 85 | 98
  Maintenance week 56, ECOG 2, n=194, 211 | 2 | 2
  Maintenance week 56, ECOG 3, n=194, 211 | 0 | 0
  Maintenance week 56, ECOG 4-5, n=194, 211 | 0 | 0
  Withdrawal from IP, ECOG 0, n=109, 92 | 44 | 38
  Withdrawal from IP, ECOG 1, n=109, 92 | 50 | 40
  Withdrawal from IP, ECOG 2, n=109, 92 | 12 | 11
  Withdrawal from IP, ECOG 3, n=109, 92 | 2 | 1
  Withdrawal from IP, ECOG 4-5, n=109, 92 | 1 | 2
  Last assessment on therapy, ECOG 0, n=334, 348 | 153 | 154
  Last assessment on therapy, ECOG 1, n=334, 348 | 158 | 165
  Last assessment on therapy, ECOG 2, n=334, 348 | 19 | 22
  Last assessment on therapy, ECOG 3, n=334, 348 | 3 | 5
  Last assessment on therapy, ECOG 4-5, n=334, 348 | 1 | 2

18. Secondary Outcome: Change From Baseline in Quality of Life Status as Assessed by the Functional Assessement of Cancer Therapy-Head and Neck (FACT-H&N) Questionnaire
Description: Change from Baseline in quality of life status was assessed using the FACT-H&N questionnaire, which is designed to measure multidimensional quality of life in participants with head and neck cancer. Change from Baseline was analyzed using parametric analysis of covariance (with the Baseline value as a covariate). The FACT-H&N questionnaire contains 39 items (27 general questions and 12 head and neck cancer-specific items) covering 4 dimensions and 1 subscale: physical well-being, social/family well-being, emotional well-being, functional well-being, and a head and neck cancer subscale. Possible subscale scores range from 0 to 36. Higher scores represent better quality of life. Data were adjusted for participant-reported quality of life scores at Baseline.
Time Frame: From randomization until the last follow-up/withdrawal visit (up to 62 study weeks)
Population: Safety Population. Only those participants who had a Baseline and post-Baseline score at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 171 | 189
scores on a scale
  Physical Well-being, n=171, 188 | 0.4 (0.33) | -0.1 (0.31)
  Social/Family Well-being, n=171, 189 | -0.3 (0.36) | -1.7 (0.34)
  Emotional Well-being, n=169, 187 | 1.0 (0.27) | 0.0 (0.26)
  Functional Well-being, n=168, 188 | 0.9 (0.39) | -0.4 (0.37)
  Head and Neck Cancer subscale, n=168, 189 | -1.2 (0.43) | -1.7 (0.40)

19. Secondary Outcome: Change From Baseline in Quality of Life Status as Assessed by the EuroQol-5D (EQ-5D) Scale
Description: Change from Baseline in quality of life status was assessed using the EQ-5D scale, a 5-item health status measure and a visual analog rating scale. Change from Baseline was analyzed using parametric analysis of covariance (with the Baseline value as a covariate). The EQ-5D is a generic measure of self-reported health outcomes that is applicable to a wide range of health conditions and treatments. The EQ-5D covers health status in 5 domains (3 questions each): mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each item is scored as follows: 1, no problems; 2, some moderate problems; 3, extreme problems. The possible EQ-5D index utility values range from 0.594 to 1, and the thermometer score ranges from 0 to 100. Higher scores represent better quality of life. Data were adjusted for participant-reported quality of life scores at Baseline.
Time Frame: From randomization until the last follow-up/withdrawal visit (up to 62 study weeks)
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 173 | 187
scores on a scale
  Utility score, n=172, 186 | 0.1 (0.01) | 0.0 (0.01)
  Thermometer score, n=173, 197 | 5.5 (1.29) | 3.2 (1.25)

20. Secondary Outcome: Number of Participants With the Indicated Biomarker Expression Status
Description: Biomarkers (which influence clinical response) assessed from tumor tissues included P16, Human Papilloma virus (HPV), and Epidermal Growth Factor Receptor (EGFR)/Epidermal Growth Factor Receptor 1 (ErbB1). Biomarker expression is presented as positive, negative, or unknown. Participants in the ErbB1-positive category include those with results of positive or strongly positive.
Time Frame: Baseline (BL; within 8 weeks prior to randomization [Day 1]) (up to Study Week 1)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 342 | 346
Participants
  P16, Positive | 42 | 48
  P16, Negative | 282 | 271
  P16, Unknown | 18 | 27
  Overall HPV, Positive | 21 | 23
  Overall HPV, Negative | 284 | 276
  Overall HPV, Unknown | 37 | 47
  ErbB1, Positive | 330 | 338
  ErbB1, Negative | 12 | 8

21. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Left Ventricular Ejection Fraction (LVEF) Change From Baseline
Description: LVEF is the measurement of how much blood is being pumped out of the left ventricle of the heart with each contraction. LVEF was assessed using echocardiogram (ECHO: a test of the action of the heart using ultrasound waves to produce a visual display, for the diagnosis or monitoring of heart disease ) and multigated acqusition scans (MUGA scan: a noninvasive diagnostic test used to evaluate the pumping function of the ventricles). Data from the ECHO and MUGA scans were combined, and the absolute change from Baseline (Abs) data are presented according to the following categories: No change or any increase, 0-<10% decrease, 10-19% decrease, >=20% decrease, >=10% decrease and >=the Lower Limit of Normal (LLN), >=10% decrease and below LLN, >=20% decrease and >=LLN, or >=20% decrease and below LLN. The relative percent change from Baseline (Rel) data are presented according to the following categories: >=20% decrease and >=LLN and >=20% decrease and below LLN.
Time Frame: From the end of the CRT until the last follow-up visit (average of 141 study weeks)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib 1500 mg
Number analyzed (Participants) | 309 | 311
Participants
  Abs, No change/any increase | 102 | 90
  Abs, >0 to <10% decrease | 138 | 131
  Abs, 10 to 19% decrease | 65 | 80
  Abs, >=20% decrease | 4 | 10
  Abs, >=10% decrease and >=LLN | 62 | 69
  Abs, >=10% decrease and below LLN | 7 | 21
  Abs, >=20% decrease and >=LLN | 3 | 5
  Abs, >=20% decrease and below LLN | 1 | 5
  Rel, >=20% decrease and >=LLN | 22 | 18
  Rel, >=20% decrease and below LLN | 3 | 14

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until the follow up of treatment (average of 141 study weeks).
Description: SAEs and non-serious AEs were reported for members of the Safety Population, comprised of all participants who were randomized and took at least one dose of study medication. Participants randomized to placebo who received >=1 dose of lapatinib in error were included in the lapatinib arm.
Arm/Group | Placebo | Lapatinib 1500 mg
Serious Adverse Events (participants affected / at risk) | 133/336 | 169/349
Other Adverse Events (participants affected / at risk) | 321/336 | 337/349
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=336) | Lapatinib 1500 mg (N=349)
Lymphopenia (Blood and lymphatic system disorders) | 17 | 18
Neutropenia (Blood and lymphatic system disorders) | 10 | 10
Anaemia (Blood and lymphatic system disorders) | 2 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 5
Leukopenia (Blood and lymphatic system disorders) | 5 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Haematotoxicity (Blood and lymphatic system disorders) | 0 | 1
Mucosal inflammation (General disorders) | 9 | 17
Pyrexia (General disorders) | 5 | 6
General physical health deterioration (General disorders) | 6 | 4
Asthenia (General disorders) | 3 | 4
Death (General disorders) | 1 | 4
Fatigue (General disorders) | 2 | 2
Impaired healing (General disorders) | 1 | 1
Malaise (General disorders) | 2 | 0
Medical device complication (General disorders) | 1 | 1
Catheter site discharge (General disorders) | 1 | 0
Catheter site related reaction (General disorders) | 0 | 1
Disease progression (General disorders) | 0 | 1
Face oedema (General disorders) | 0 | 1
Mucosal induration (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Performance status decreased (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 8 | 12
Dysphagia (Gastrointestinal disorders) | 5 | 11
Nausea (Gastrointestinal disorders) | 3 | 7
Diarrhoea (Gastrointestinal disorders) | 3 | 6
Stomatitis (Gastrointestinal disorders) | 5 | 4
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 3
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 2
Oral pain (Gastrointestinal disorders) | 1 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastrooesophagitis (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Oesophageal fistula (Gastrointestinal disorders) | 1 | 0
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Stomatitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 12
Dehydration (Metabolism and nutrition disorders) | 5 | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 5
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3
Malnutrition (Metabolism and nutrition disorders) | 2 | 4
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3
Feeding disorder (Metabolism and nutrition disorders) | 0 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 6
Sepsis (Infections and infestations) | 2 | 4
Wound infection (Infections and infestations) | 0 | 3
Bronchopneumonia (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Lung abscess (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 1 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 1
Oral infection (Infections and infestations) | 0 | 2
Abscess limb (Infections and infestations) | 0 | 1
Abscess neck (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Blister infected (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Paraoesophageal abscess (Infections and infestations) | 0 | 1
Parotid abscess (Infections and infestations) | 1 | 0
Perichondritis (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis syndrome (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Superinfection (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Ejection fraction decreased (Investigations) | 3 | 10
Blood creatinine increased (Investigations) | 2 | 5
Hepatic enzyme increased (Investigations) | 2 | 3
Weight decreased (Investigations) | 1 | 4
Alanine aminotransferase increased (Investigations) | 3 | 1
Blood uric acid increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 1
Alanine aminotransferase abnormal (Investigations) | 0 | 1
Blood bilirubin abnormal (Investigations) | 0 | 1
Calcium ionised decreased (Investigations) | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1
Electrocardiogram change (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Osteoradionecrosis (Injury, poisoning and procedural complications) | 6 | 1
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1 | 3
Radiation mucositis (Injury, poisoning and procedural complications) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 1
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Feeding tube complication (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Foreign body (Injury, poisoning and procedural complications) | 1 | 0
Implant tissue necrosis (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Radiation sickness syndrome (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Syncope (Nervous system disorders) | 2 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 2
Ataxia (Nervous system disorders) | 0 | 1
Brain hypoxia (Nervous system disorders) | 1 | 0
Brain injury (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1
Paralysis (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 3 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 1
Intracardiac mass (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Ventricular hypokinesia (Cardiac disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oral fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 4
Skin reaction (Skin and subcutaneous tissue disorders) | 3 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pemphigus (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 2 | 0
Arterial rupture (Vascular disorders) | 1 | 0
Arterial thrombosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 3
Renal failure acute (Renal and urinary disorders) | 3 | 0
Renal impairment (Renal and urinary disorders) | 1 | 2
Depression (Psychiatric disorders) | 1 | 2
Completed suicide (Psychiatric disorders) | 1 | 1
Suicide attempt (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Neurosensory hypoacusis (Ear and labyrinth disorders) | 0 | 1
Aplasia (Congenital, familial and genetic disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 1
Hepatitis E (Infections and infestations) | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=336) | Lapatinib 1500 mg (N=349)
Alanine aminotransferase increased (Investigations) | 31 | 30
Aspartate aminotransferase increased (Investigations) | 28 | 33
Blood creatinine increased (Investigations) | 33 | 44
Creatinine renal clearance decreased (Investigations) | 17 | 27
Haemoglobin decreased (Investigations) | 29 | 33
Lymphocyte count decreased (Investigations) | 18 | 20
Weight decreased (Investigations) | 64 | 90
White blood cell count decreased (Investigations) | 23 | 30
Anaemia (Blood and lymphatic system disorders) | 61 | 77
Leukopenia (Blood and lymphatic system disorders) | 99 | 83
Lymphopenia (Blood and lymphatic system disorders) | 75 | 87
Neutropenia (Blood and lymphatic system disorders) | 77 | 70
Thrombocytopenia (Blood and lymphatic system disorders) | 25 | 24
Asthenia (General disorders) | 45 | 59
Fatigue (General disorders) | 36 | 41
Mucosal inflammation (General disorders) | 208 | 220
Pyrexia (General disorders) | 60 | 63
Constipation (Gastrointestinal disorders) | 74 | 60
Diarrhoea (Gastrointestinal disorders) | 41 | 147
Dry mouth (Gastrointestinal disorders) | 131 | 148
Dyspepsia (Gastrointestinal disorders) | 21 | 30
Dysphagia (Gastrointestinal disorders) | 113 | 125
Nausea (Gastrointestinal disorders) | 150 | 181
Odynophagia (Gastrointestinal disorders) | 34 | 41
Oral pain (Gastrointestinal disorders) | 35 | 25
Stomatitis (Gastrointestinal disorders) | 50 | 50
Vomiting (Gastrointestinal disorders) | 115 | 154
Cough (Respiratory, thoracic and mediastinal disorders) | 37 | 45
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 21 | 23
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 67 | 45
Productive cough (Respiratory, thoracic and mediastinal disorders) | 36 | 25
Decreased appetite (Metabolism and nutrition disorders) | 69 | 62
Hypokalaemia (Metabolism and nutrition disorders) | 28 | 42
Hyponatraemia (Metabolism and nutrition disorders) | 25 | 33
Dysgeusia (Nervous system disorders) | 45 | 31
Headache (Nervous system disorders) | 28 | 20
Insomnia (Psychiatric disorders) | 20 | 17
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 23 | 15
Neck pain (Musculoskeletal and connective tissue disorders) | 28 | 20
Oral candidiasis (Infections and infestations) | 22 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 23
Rash (Skin and subcutaneous tissue disorders) | 101 | 167
Skin reaction (Skin and subcutaneous tissue disorders) | 37 | 41
Radiation mucositis (Injury, poisoning and procedural complications) | 19 | 13
Radiation skin injury (Injury, poisoning and procedural complications) | 79 | 55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.